CLINICAL TRIAL: NCT06153277
Title: Does Edema After Knee Arthroplasty Affect the Adjustment of TENS Amplitude
Brief Title: Does Edema Affect the Adjustment of TENS Amplitude
Status: Recruiting | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aynur Başaran, Proffessor Dr, MD, Karamanoğlu Mehmetbey University
Other Study IDs: 09-2023/01
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Edema Leg; Pain
Keywords: Transcutaneous electrical nerve stimulation; Amplitude adjustment; Arthroplasty
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pre-post clinical trial is to compare the amplitude settings of three different frequency TENS modes (Conventional TENS, LF TENS, HF TENS) in patients who had undergone total knee arthroplasty, both with the preoperative state and with the contralateral knee. The main question it aims to answer is: Can the electrical resistance of edematous tissue be affected and change the TENS amplitude setting? Participants will be evaluated before and after surgery. For each TENS modulation the amplitude at which tingling is felt, the current is clearly felt, and is maximum tolerated and/or muscle contraction occurred, will be documented. TENS amplitudes for all three TENS modes will be compared, both with the preoperative state and with the contralateral knee.

DETAILED DESCRIPTION:
Transcutaneous Electrical Nerve Stimulation (TENS) is used for the treatment of various acute and chronic pain conditions. It has been shown to increase participation by providing pain control in the rehabilitation of patients undergoing surgery. Evidence is accumulating that it improves patient comfort and reduces the use of analgesic medication in the early postoperative period, so TENS is included in postoperative pain management guidelines.

On the other hand, peripheral blocks have become the preferred method of anesthesia in order to avoid the complications of general anesthesia. When adjusting TENS amplitude for postoperative pain control in these patients, either low amplitudes are preferred or for the amplitude adjustment as a reference, the contralateral side without block is used.

Cautious application is recommended in patients with sensory impairment, impaired cognitive functions, and pediatric patients. In such cases, it is preferable to use TENS at low amplitudes to avoid complications in daily practice. However, using the contralateral extremity as a reference may cause undesirable results as the electrical resistance of the edematous tissue may change.

In this study, it was aimed to compare the amplitude settings of three different frequency TENS modes (Conventional TENS, LF TENS, HF TENS) in patients who had undergone total knee arthroplasty, both in the preoperative state and with the contralateral knee.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Patients undergoing unilateral total knee arthroplasty

Exclusion Criteria:

* Patients with scars in any of both knee areas
* Patients who have previously had surgery on the control leg
* Patients undergoing surgery due to trauma or cancer
* Patients with sensory impairments
* Patients with excessive effusion and edema in the knee joints before the surgery (eg. Inflammatory arthropathy, gonarthrosis exacerbation, etc.)
* Mental impairment, or poor general health status that would interfere with assessments during TENS application.
* Any contraindication for TENS (allergy to the TENS electrodes, skin conditions or skin sensation impairment in the areas where the electrodes will be placed, pacemaker or other implanted electrical device, epilepsy, pregnancy)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Karaman Training and Research Hospital Orthopedics and Traumatology Polyclinic and were planned for unilateral knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The difference in amplitudes of the conventional TENS mode between pre- and post-arthroplasty measurements | 2-3 days
  Univariate statistical analyses will be performed to calculate differences in amplitudes of the conventional TENS mode between pre- and post-arthroplasty measurements on both knees and between knees
The difference in amplitudes of the high frequency TENS mode between pre- and post-arthroplasty measurements | 2-3 days
  Univariate statistical analyses will be performed to calculate differences in amplitudes of the high frequency TENS mode between pre- and post-arthroplasty measurements on both knees and between knees
The difference in amplitudes of the low frequency TENS mode between pre- and post-arthroplasty measurements | 2-3 days
  Univariate statistical analyses will be performed to calculate differences in amplitudes of the low frequency TENS mode between pre- and post-arthroplasty measurements on both knees and between knees

SECONDARY OUTCOMES:
The effect of the amount of edema on the amplitudes of TENS modes | 2-3 days
  Primary study results found to be significant in univariate analysis will be checked for correlation with the amount of edema in the operated knee
The effect of the type of anesthesia applied on the amplitudes of TENS modes | 203 days
  Primary study results found to be significant in univariate analysis will be tested with post-hoc analysis whether the type of anesthesia applied has any effect

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Basaran, MD,Prof, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)